CLINICAL TRIAL: NCT03874832
Title: A Randomized, Open-Label, Crossover Study to Evaluate the PK, Bioavailability, Dose Proportionality, Safety, and Tolerability of Single Doses of STS101, DHE Mesylate IM Injection and DHE Mesylate Nasal Spray in Healthy Adult Subjects
Brief Title: A Phase I Study to Study the PK and Safety of Single Doses of STS101, DHE Injection and Nasal Spray in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Satsuma Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STS101-001
Record Dates: First submitted 2019-03-07; First posted 2019-03-14 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Migraine With Aura; Migraine Without Aura; Migraine
Keywords: dihydroergotamine; dihydroergotamine mesylate; migraine
MeSH Terms: conditions — Migraine with Aura; Migraine without Aura; Migraine Disorders | interventions — Dihydroergotamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- STS101 1.5 mg (Experimental): STS101 (dihydroergotamine nasal powder), 1.5 mg
  Interventions: Drug: Dihydroergotamine
- STS101 3.0 mg (Experimental): STS101 (dihydroergotamine nasal powder), 3.0 mg
  Interventions: Drug: Dihydroergotamine
- STS101 6.0 mg (Experimental): STS101 (dihydroergotamine nasal powder), 6.0 mg
  Interventions: Drug: Dihydroergotamine
- DHE intramuscular injection (Active Comparator): Dihydroergotamine mesylate
  Interventions: Drug: Dihydroergotamine
- DHE nasal spray (Active Comparator): Dihydroergotamine mesylate
  Interventions: Drug: Dihydroergotamine

INTERVENTIONS:
Drug: Dihydroergotamine — Dihydroergotamine is a semi-synthetic derivative of ergotamine tartrate.
  Other Names: Dihydroergotamine Mesylate

SUMMARY:
Single-center, single-dose, open-label, 2-part, 3-period crossover (in each part), pharmacokinetic and safety study.

DETAILED DESCRIPTION:
Phase 1, open-label, 2-part, single-dose pharmacokinetic and safety study of STS101 in healthy subjects. Part 1 was designed to identify a dose level of STS101 for administration in Part 2. Subjects in Part 1 received 3 ascending doses of STS101 in a 3-period crossover manner. During Part 2, subjects received the dose of STS101 selected from Part 1, 1.0 mg DHE mesylate IM injection, and 2 mg DHE mesylate nasal spray in a randomized, 3 period crossover manner.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years of age at the time of enrollment.
* Signed the informed consent document.
* Subject judged to be healthy by a qualified physician

Exclusion Criteria:

* Abnormal physical findings of clinical significance at the screening examination
* Significant abnormal laboratory values at the Screening Visit.
* Clinically significant symptoms or conditions that may have placed the subject at an unacceptable risk as a participant in the trial, or that may have interfered with the absorption, distribution, metabolism or excretion of the IMP.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
STS101 Dose Selection - Part 1 | Pre-dose through 48 hours post-dose
  To select a dose level of STS101 for further evaluation in Part 2
DHE Relative Bioavailability - Part 2 | Pre-dose through 48 hours post-dose
  To assess the relative bioavailability of dihydroergotamine following a single dose of STS101 at the dose level selected in Part 1 compared to a single dose of 1 mg DHE administered by intramuscular injection and 2 mg DHE administered as nasal spray

SECONDARY OUTCOMES:
DHE Area Under the Curve [AUC] - Part 1 | Pre-dose through 48 hours post-dose
  To describe the pharmacokinetic profile based on the AUC of dihydroergotamine following single dose administration of 1.5 mg, 3.0 mg and 6.0 mg of STS101
8'OH-DHE Area Under the Curve [AUC] - Part 1 | Pre-dose through 48 hours post-dose
  To describe the pharmacokinetic profile based on the AUC of 8'hydroxydihydroergotamine (8'OH-DHE) following single dose administration of 1.5 mg, 3.0 mg and 6.0 mg of STS101
Serious Adverse Events - Parts 1 & 2 | Pre-dose through 48 hours post-dose
  To assess the safety profile through examination of serious adverse events of single doses of STS101; 1 mg DHE administered by intramuscular injection, and 2 mg DHE administered as nasal spray
Treatment-Related Adverse Events - Parts 1 & 2 | Pre-dose through 48 hours post-dose
  To assess the safety profile through examination of treatment-related adverse events of single doses of STS101; 1 mg DHE administered by intramuscular injection, and 2 mg DHE administered as nasal spray

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Levy, MD, PhD, Principal Investigator — Quotient Sciences Miami Inc.
Locations (1):
- Quotient Sciences Miami Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Albrecht D, Iwashima M, Dillon D, Harris S, Levy J. A Phase 1, Randomized, Open-Label, Safety, Tolerability, and Comparative Bioavailability Study of Intranasal Dihydroergotamine Powder (STS101), Intramuscular Dihydroergotamine Mesylate, and Intranasal DHE Mesylate Spray in Healthy Adult Subjects. Headache. 2020 Apr;60(4):701-712. doi: 10.1111/head.13737. Epub 2020 Jan 27. PMID 31985049